CLINICAL TRIAL: NCT04847557
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study Comparing the Efficacy and Safety of Tirzepatide Versus Placebo in Patients With Heart Failure With Preserved Ejection Fraction and Obesity (SUMMIT)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF) and Obesity: The SUMMIT Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17757; I8F-MC-GPID (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-02-26; First posted 2021-04-19 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Heart Failure with Preserved Ejection Fraction (HFpEF)
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants received a starting dose of 2.5 milligrams (mg) tirzepatide administered subcutaneously (SC) once weekly (QW) and escalated by 2.5 mg every 4 weeks to a maximum of 15 mg QW or maximum tolerated dose (MTD) tolerated by the participant (5 mg QW or 10 mg QW).
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received placebo administered SC QW.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of Tirzepatide (LY3298176) in participants with heart failure with preserved ejection fraction and obesity.

DETAILED DESCRIPTION:
The study will continue until approximately 52 weeks after the last participant is randomized. The maximum duration of an individual's participation is estimated to be ~120 weeks and will depend on duration of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of stable heart failure (NYHA class II-IV) and left ventricular ejection fraction (LVEF) ≥50%
* Elevated NT-proBNP (N-terminal pro B-type natriuretic peptide) > 200 picogram/milliliter (pg/ml) for participants without atrial fibrillation (AF), or >600 pg/ml for participants with AF, Structural heart disease (Left atrial enlargement) or Elevated left ventricular filling pressure
* Estimated glomerular filtration rate (eGFR) <70 milliliter (ml)/minute (min)/1.73m² at screening, or HF decompensation within 12 months of screening,
* Stable dose of heart failure medications within 4 weeks of screening
* Body mass index (BMI) ≥30 kilograms per meter squared (kg/m²)
* 6MWD 100-425 meters
* KCCQ CSS ≤80

Exclusion Criteria:

* Have had a major cardiovascular event within the last 90 days of screening
* Have had acute decompensated heart failure within 4 weeks of screening
* Have non cardiac causes of functional impairment such as pulmonary arterial hypertension (PAH), severe chronic obstructive pulmonary disease (COPD), anemia, thyroid disease, musculoskeletal disease or orthopedic conditions
* Presence of cardiac amyloidosis, cardiac accumulation disease, cardiomyopathy and severe valvular heart disease
* HbA1c ≥9.5% or uncontrolled diabetes
* History of proliferative diabetic retinopathy or diabetic maculopathy
* Have a history of pancreatitis
* eGFR <15 mL/min/1.73 m² or requiring dialysis at screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (146):
- United States (54):
  - Heart Center Research, Huntsville, Alabama
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Valley Clinical Trials, Inc., Covina, California
  - Amicis Research Center, Granada Hills, California
  - University of California San Diego - La Jolla, La Jolla, California
  - Valley Clinical Trials, Inc., Northridge, California
  - The Lundquist Institute, Torrance, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Clearwater, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Largo, Florida
  - Infinite Clinical Research, Miami, Florida
  - Ocala Caridovascular Research, Ocala, Florida
  - Clearwater Cardiovascular & Interventional Consultants M.D., P.A., Safety Harbor, Florida
  - East Coast Institute for Research - St. Augustine, Saint Augustine, Florida
  - Morehouse School Of Medicine, Atlanta, Georgia
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Northwest Heart Clinical Research, Arlington Heights, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Cardiovascular Research of Northwest Indiana, Munster, Indiana
  - Midwest Heart & Vascular Specialists, Overland Park, Kansas
  - Grace Research - Bossier, Bossier City, Louisiana
  - The Heart Clinic - Hammond, Hammond, Louisiana
  - Grace Research - Shreveport, Shreveport, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - McLaren Bay Region, Bay City, Michigan
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - The Heart House, Haddon Heights, New Jersey
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Erie County Medical Center, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - Saratoga Cardiology Associates, Saratoga Springs, New York
  - Stony Brook University, Stony Brook, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Aultman Hospital Research, Canton, Ohio
  - Rama Research, Marion, Ohio
  - Hightower Clinical Trial Services, Oklahoma City, Oklahoma
  - Hillsboro Cardiology, Hillsboro, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Clinical Trials, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Apex Research Foundation, Jackson, Tennessee
  - DiscoveResearch, Beaumont, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Intermountain Medical Center, Murray, Utah
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
- Argentina (17):
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires, Buenos Aires F.D.
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Air
  - CIPREC, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - CEMEDIC, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Instituto de Cardiología "Juana F. Cabral", Corrientes
  - Centro de Investigaciones Clinicas Instituto del Corazon (CICIC), Córdoba
  - Hospital de Alta Complejidad "Pte. Juan Domingo Perón", Formosa
  - Centro Cardiovascular Salta, Salta
  - Instituto Cardiovascular San Luis, San Luis
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Brazil (11):
  - Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Angelina Caron, Campina Grande do Sul, Paraná
  - Centro de Pesquisa Clinica do Coracao, Aracaju, Sergipe
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Loema Instituto de Pesquisa Clinica, Campinas, São Paulo
  - CAPED Centro Avancado Pesquisa e Diagnostica, Ribeirão Preto, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- China (21):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Lanzhou university second hospital, Lanzhou, Gansu
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan University Medical College - Hubei Zhongshan Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - 1st Hospital affiliate to Baotou medical college, Baotou, Inner Mongolia
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - China-Japan Union Hospital, Changchun, Jilin
  - The first affiliated hospital of dalian medical university, Dalian, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
- India (10):
  - CIMS Hospital - Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Medanta The Medicity, Gurugramam, Haryana
  - Narayana Institute of Cardiac Sciences, Bangalore, Karnataka
  - King Edward Memorial Hospital & Seth Gordhandas Sunderdas Medical College, Mumbai, Maharashtra
  - Government Medical College And Hospital - Nagpur, Nagpur, Maharashtra
  - Central India Cardiology and Research Institute, Nagpur, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Centre, New Delhi, National Capital Territory of Delhi
  - AIG Hospitals, Hyderabad, Telangana
- Israel (11):
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Hillel Yaffe Medical Center, Hadera, Northern District
  - Rambam Health Care Campus, Haifa, Northern District
  - Galilee Medical Center, Nahariya, Northern District
  - Barzilai Medical Center, Ashkelon, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Mexico (7):
  - CIMAB SA de CV, Torreón, Coahuila
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Hospital Cardiologica Aguescalientes, Aguascalientes
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
- Puerto Rico (2):
  - Clinical Research Center - Universidad Central del Caribe (CRC - UCC), Bayamón
  - Research and Cardiovascular Corp., Ponce
- Russia (6):
  - Ivanovo Regional Healthcare Institution Cardiology Dispensary, Ivanovo, Ivanovo Oblast
  - Russian Cardiology Research and Production Complex, Moscow, Moscow
  - Russian Medical Academy of Postgraduate Education, Moscow, Moscow
  - Ryazan Regional Clinical Cardiological Dispensary, Ryazan, Ryazan Oblast
  - Astarta Clinic, Saint Petersburg, Sankt-Peterburg
  - Izhevsk City Clinical Hospital Number 9, Izhevsk, Udmurtiya Republic
- Taiwan (7):
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Mackay Memorial Hospital-Hsinchu, Hsinchu
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Packer M, Zile MR, Kramer CM, DiMaria JM, Baum SJ, Litwin SE, Murakami M, Zhou C, Ou Y, Koeneman L, Borlaug BA; SUMMIT Trial Study Group. Influence of Type 2 Diabetes on the Effects of Tirzepatide in Patients With Heart Failure and a Preserved Ejection Fraction With Obesity: A Prespecified Stratification-Based Analysis. J Am Coll Cardiol. 2025 Sep 9;86(10):696-707. doi: 10.1016/j.jacc.2025.06.058. PMID 40903131
- [Derived] Borlaug BA, Zile MR, Kramer CM, Ye W, Ou Y, Hurt K, Murakami M, Packer M; SUMMIT Trial Study Group. Impact of Body Mass Index, Central Adiposity, and Weight Loss on the Benefits of Tirzepatide in HFpEF: The SUMMIT Trial. J Am Coll Cardiol. 2025 Jul 29;86(4):242-255. doi: 10.1016/j.jacc.2025.04.059. PMID 40701669
- [Derived] Packer M, Zile MR, Kramer CM, Murakami M, Ou Y, Borlaug BA; SUMMIT Trial Study Group. Interplay of Chronic Kidney Disease and the Effects of Tirzepatide in Patients With Heart Failure, Preserved Ejection Fraction, and Obesity: The SUMMIT Trial. J Am Coll Cardiol. 2025 May 13;85(18):1721-1735. doi: 10.1016/j.jacc.2025.03.009. Epub 2025 Mar 31. PMID 40162940
- [Derived] Kramer CM, Borlaug BA, Zile MR, Ruff D, DiMaria JM, Menon V, Ou Y, Zarante AM, Hurt KC, Murakami M, Packer M; SUMMIT Trial Study Group. Tirzepatide Reduces LV Mass and Paracardiac Adipose Tissue in Obesity-Related Heart Failure: SUMMIT CMR Substudy. J Am Coll Cardiol. 2025 Feb 25;85(7):699-706. doi: 10.1016/j.jacc.2024.11.001. Epub 2024 Nov 18. PMID 39566869
- [Derived] Zile MR, Borlaug BA, Kramer CM, Baum SJ, Litwin SE, Menon V, Ou Y, Weerakkody GJ, Hurt KC, Kanu C, Murakami M, Packer M; SUMMIT Trial Study Group. Effects of Tirzepatide on the Clinical Trajectory of Patients With Heart Failure, Preserved Ejection Fraction, and Obesity. Circulation. 2025 Mar 11;151(10):656-668. doi: 10.1161/CIRCULATIONAHA.124.072679. Epub 2024 Nov 18. PMID 39556714
- [Derived] Packer M, Zile MR, Kramer CM, Baum SJ, Litwin SE, Menon V, Ge J, Weerakkody GJ, Ou Y, Bunck MC, Hurt KC, Murakami M, Borlaug BA; SUMMIT Trial Study Group. Tirzepatide for Heart Failure with Preserved Ejection Fraction and Obesity. N Engl J Med. 2025 Jan 30;392(5):427-437. doi: 10.1056/NEJMoa2410027. Epub 2024 Nov 16. PMID 39555826
- [Derived] Borlaug BA, Zile MR, Kramer CM, Baum SJ, Hurt K, Litwin SE, Murakami M, Ou Y, Upadhyay N, Packer M. Effects of tirzepatide on circulatory overload and end-organ damage in heart failure with preserved ejection fraction and obesity: a secondary analysis of the SUMMIT trial. Nat Med. 2025 Feb;31(2):544-551. doi: 10.1038/s41591-024-03374-z. Epub 2024 Nov 17. PMID 39551891
- See also: A Study of Tirzepatide (LY3298176) in Participants With Heart Failure With Preserved Ejection Fraction and Obesity (SUMMIT) — https://trials.lillytrialguide.com/en-US/trial/4deAJHqkMfFYm9JjtgeqTl

RESULTS

PARTICIPANT FLOW:
Groups:
- Tirzepatide - MTD: Participants received a starting dose of 2.5 milligrams (mg) tirzepatide administered subcutaneously (SC) once weekly (QW) and escalated by 2.5 mg every 4 weeks to a maximum of 15 mg QW or maximum tolerated dose (MTD) tolerated by the participant (5 mg QW or 10 mg QW).
Period: Overall Study
Arm/Group | Tirzepatide - MTD | Placebo
Started | 364 | 367
Received At Least One Dose of Study Drug | 364 | 367
Completed | 332 | 331
Not Completed | 32 | 36
Not completed — Adverse Event | 1 | 0
Not completed — Death | 19 | 15
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 8 | 14

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Tirzepatide - MTD: Participants received a starting dose of 2.5 mg tirzepatide administered SC QW and escalated by 2.5 mg every 4 weeks to a maximum of 15 mg QW or MTD tolerated by the participant (5 mg QW or 10 mg QW).
- Total: Total of all reporting groups
Arm/Group | Tirzepatide - MTD | Placebo | Total
Number analyzed (Participants) | 364 | 367 | 731
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.50 (10.53) | 65.00 (10.87) | 65.20 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 193 | 393
  Male | 164 | 174 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 195 | 205 | 400
  Not Hispanic or Latino | 164 | 159 | 323
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 23 | 47
  Asian | 58 | 73 | 131
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 22 | 14 | 36
  White | 256 | 256 | 512
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 101 | 103 | 204
  Brazil | 51 | 54 | 105
  China | 25 | 30 | 55
  India | 9 | 11 | 20
  Israel | 17 | 21 | 38
  Mexico | 41 | 40 | 81
  Russia | 13 | 8 | 21
  Taiwan | 24 | 32 | 56
  United States | 83 | 68 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS)
Description: The KCCQ is a 23-item, participant self-administered questionnaire that assesses impacts of heart failure "over the past 2 weeks" on the following 7 domains:
  * Physical Limitation (6)
  * Symptom Stability (1)
  * Symptom Frequency (4)
  * Symptom Burden (3)
  * Self-Efficacy (2)
  * Quality of Life (3)
  * Social Limitation (4)
  Each of the 23 individual items are answered on Likert scales of varying lengths (5, 6, or 7-point scales).
  KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are obtained by averaging the associated individual items and transforming the score to a 0 to 100 range. Higher scores indicate better health status.
  Least Square (LS) mean was determined using ANCOVA model with Baseline + HF Decompensation Within 12 Months of Screening + T2DM Status + Baseline BMI group (<35, >=35 kg/m2) + Treatment (Type III sum of squares) as variables .
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 301 | 313
Score on a scale | 19.51 (1.24) | 12.68 (1.25)
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; p < 0.001, Stratified Wilcoxon; Stratified Wilcoxon test used to control for stratification factors of HF decompensation within 12 months of screening,diagnosed T2DM & baseline BMI; Median Difference (Net) = 6.9, 95% CI 2-sided [3.3 to 10.6] — The Hodges-Lehmann estimate for the median difference and 95% CIs was reported

2. Primary Outcome: First Occurrence of the Composite Endpoint of Heart Failure (HF) Outcomes
Description: Clinical Endpoint Committe confirmed Occurrences of CV outcomes were reported here. HF outcomes consisted of cardiovascular death and HF events.
  The HF events were defined as worsening clinical symptoms or signs related to HF, which are meaningful to the participant and require intensification of treatment characterized by 1 or more of the following:
  * hospitalization for heart failure regardless of duration or treatment received
  * use of intravenous drug, usually an intravenous diuretic, but may include intravenous vasodilators or positive inotropic drugs, or
  * augmentation or increase in oral diuretic therapy.
Time Frame: Baseline Up To 160 weeks
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Number of events
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Number of events | 36 | 56
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Heart Failure Outcomes; Test type: Superiority; p = 0.026, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.41 to 0.95]

3. Secondary Outcome: Change From Baseline in Exercise Capacity as Measured by 6-Minute Walk Distance (6MWD)
Description: Participants performed an exercise capacity assessment using the 6-Minute Walk Test (6MWT) and the distance covered (6MWD) was assessed in meters. The 6MWT was performed indoors on a straight, flat, hard surface that is at least 30 meters in length. The greater distance walked meant better physical capacity.
  LS Mean was determined using ANCOVA model with Baseline + HF Decompensation Within 12 Months of Screening + T2DM Status + Baseline BMI group (<35, >=35 kg/m2) + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome,
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 326 | 314
meters | 26.04 (3.81) | 10.10 (3.94)
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; p < 0.001, Stratified Wilcoxon; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = 18.3, 95% CI 2-sided [9.9 to 26.7] — The Hodges-Lehmann estimate for the median difference and 95% CIs was reported

4. Secondary Outcome: Percent Change From Baseline in Body Weight
Description: Percent change in bodyweight was reported. LS mean was determined using ANCOVA model with Baseline + HF Decompensation Within 12 Months of Screening + T2DM Status + Baseline BMI group (<35, >=35 kg/m2) + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 331 | 333
Percent change | -13.85 (0.43) | -2.24 (0.46)
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -11.62, 95% CI 2-sided [-12.85 to -10.38]

5. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP)
Description: Percent change from baseline in hsCRP was reported. LS Mean was determined using ANCOVA model with log (actual measurement/baseline) = log (baseline) + HF decompensation within 12 months of screening + T2DM status + baseline BMI group (<35, >=35 kg/m2) + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 305 | 298
Percent change | -38.76 (4.47) | -5.88 (5.25)
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -34.91, 95% CI 2-sided [-45.60 to -22.17]

6. Secondary Outcome: Win Percentage of the Hierarchical Composite Endpoint
Description: Hierarchical Composite Endpoint included time to all-cause death, number of HF events, time to first HF events, KCCQ-CSS, 6MWD.
  The winner was determined in each pair-wise comparison in the following order:
  * A delayed first occurrence of all-cause death
  * If the pair cannot be differentiated based on death, winner has fewer HF events
  * If the pair cannot be differentiated by number of HF events, winner has delayed time to occurrence of first HF event
  * If the pair still cannot be differentiated, winner has a more favorable category for change from baseline in 6MWD
  * If the pair still cannot be differentiated, winner has a more favorable category for change from baseline in KCCQ-CSS
  * Otherwise the pair will be recorded as tied.
  Reported unit is the total percent of "wins" for each treatment group from performing such a hierarchical comparison across stratification factors in the study.
Time Frame: Baseline Up To 160 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Win percentage
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Win percentage | 57.90 | 35.43
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Win Ratio = 1.63, 95% CI 2-sided [1.17 to 2.28] — The win ratio was reported as the measure of treatment effect based on the principle that each participant is compared with every other participant within each stratum in a pair-wise manner that proceeds in a hierarchical fashion

7. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class Change
Description: Percentage of participants with NYHA class change at Week 52 was reported.
Time Frame: Week 52
Population: All participant who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 328 | 327
Percentage of participants | 33.27 | 20.39
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.53 to 3.40]

8. Secondary Outcome: Number of Participants With Time to All-Cause Death
Description: All-cause mortality is death due to any cause. Number of participants with time to all-cause mortality are presented.
Time Frame: Baseline Up To 160 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Participants | 19 | 15
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.245, 95% CI 2-sided [0.633 to 2.452]

9. Secondary Outcome: Number of Participants With Time to First Occurrence of HF Events
Description: Number of participants with time to first occurrence of HF events are reported.
Time Frame: Baseline Up To 160 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Participants | 29 | 52
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.539, 95% CI 2-sided [0.342 to 0.850]

10. Secondary Outcome: Number of HF Events and All-Cause Death
Description: Number of HF events and all-cause death are reported.
Time Frame: Baseline Up To 160 Weeks.
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Events
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Events | 61 | 82
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Rate Ratio = 0.72, 95% CI 2-sided [0.46 to 1.14]

11. Secondary Outcome: Number of Recurrent HF Events
Description: Number of recurrent HF events were reported.
Time Frame: Baseline Up To 160 Weeks.
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Events
Arm/Group | Tirzepatide - MTD | Placebo
Number analyzed (Participants) | 364 | 367
Events | 44 | 68
Statistical Analysis 1: Comparison: Tirzepatide - MTD vs Placebo; Test type: Superiority; Rate Ratio = 0.62, 95% CI 2-sided [0.37 to 1.05]

ADVERSE EVENTS:
Time Frame: Baseline Up To 162 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse event analysis was planned as per the treatment regimen received.
Arm/Group | Tirzepatide - MTD | Placebo
All-Cause Mortality (participants affected / at risk) | 19/364 | 15/367
Serious Adverse Events (participants affected / at risk) | 96/364 | 94/367
Other Adverse Events (participants affected / at risk) | 221/364 | 137/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tirzepatide - MTD (N=364) | Placebo (N=367)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (7)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (3) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 7 (9) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 12 (17) | 18 (27)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 12 (18)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial bridging (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pacemaker syndrome (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 2 (2) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 6 (7)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 3 (5) | 4 (4)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/200 (1) | 0/193 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/164 (0) | 1/174 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/164 (0) | 1/174 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/200 (0) | 1/193 (2)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Prosthetic cardiac valve malfunction (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 2 (3)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Distributive shock (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide - MTD (N=364) | Placebo (N=367)
Cardiac failure (Cardiac disorders) | 11 (19) | 20 (24)
Abdominal pain upper (Gastrointestinal disorders) | 19 (24) | 7 (10)
Constipation (Gastrointestinal disorders) | 54 (78) | 22 (27)
Diarrhoea (Gastrointestinal disorders) | 65 (185) | 23 (33)
Dyspepsia (Gastrointestinal disorders) | 23 (30) | 8 (11)
Nausea (Gastrointestinal disorders) | 62 (214) | 23 (32)
Vomiting (Gastrointestinal disorders) | 38 (71) | 7 (9)
Covid-19 (Infections and infestations) | 33 (35) | 41 (45)
Urinary tract infection (Infections and infestations) | 31 (42) | 22 (25)
Decreased appetite (Metabolism and nutrition disorders) | 38 (42) | 6 (7)
Dizziness (Nervous system disorders) | 34 (81) | 18 (20)
Hypotension (Vascular disorders) | 22 (25) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04847557/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT04847557/SAP_001.pdf